CLINICAL TRIAL: NCT01088126
Title: Comparison of Linear Ablation Versus Focal Ablation of Complex Fractionated Atrial Electrograms After Pulmonary Vein Isolation in Patients With Persistent Atrial Fibrillation: A Prospective & Randomized Controlled Study
Brief Title: Linear Ablation Versus Focal Ablation of Complex Fractionated Atrial Electrograms in Persistent Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It was difficult to enrol patients.
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Young-Hoon Kim, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN09239
Record Dates: First submitted 2010-03-01; First posted 2010-03-17 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2010-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

ARMS (2):
- Focal ablation (Active Comparator): PV isolation + CFAE-targeted focal ablation
  Interventions: Procedure: radiofrequency catheter ablation
- Linear ablation (Active Comparator): PV isolation + CFAE-guided linear ablation
  Interventions: Procedure: radiofrequency catheter ablation

INTERVENTIONS:
Procedure: radiofrequency catheter ablation — radiofrequency catheter ablation, NavX system

SUMMARY:
The end point of catheter ablation at complex fractionated atrial electrograms (CFAE) was not established yet. Furthermore, incomplete CFAE ablation may have a potential to develop atrial tachyarrhythmias (AT). The investigators hypothesized that linear ablation extending the clusters of CFAE would be a better strategy than focal ablation at the individual CFAE sites.

ELIGIBILITY:
Inclusion Criteria:

* patients age 18 or greater
* persistent atrial fibrillation
* candidates for AF ablation based on AF that is symptomatic and refractory to at least one antiarrhythmic medication
* at least one episode of AF must have been documented by ECG or Holter within 12 months of randomization in the trial
* continuous anticoagulation with warfarin (INR 2-3) for >4 weeks prior to the ablation
* patients must be able and willing to provide written informed consent to participate in the clinical trial

Exclusion Criteria:

* paroxysmal or permanent atrial fibrillation
* patients with AF felt to be secondary to an obvious reversible cause
* inadequate anticoagulation as defined in the inclusion criteria
* left atrial thrombus on TEE prior to procedure
* contraindications to systemic anticoagulation with heparin or coumadin
* previously undergone atrial fibrillation ablation
* patients who are or may potentially be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
freedom from AF/AT more than 3 months after first ablation | 12 months

SECONDARY OUTCOMES:
freedom from AF/AT within 3 months following first ablation | 3 months
acute intra-procedure termination of AF | 12 months
organization of AF/conversion to AT during the ablation | 12 months
procedure time | 12 months
ablation time | 12 months
procedure-related complication | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Kim, M.D., Ph.D., Principal Investigator — Korea University
Locations (1):
- Korea University Medical Center, Seoul, South Korea